CLINICAL TRIAL: NCT00176410
Title: Statin Therapy in Asymptomatic Aortic Stenosis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Leipzig (Other)
Collaborators: Novartis (Industry)
Responsible Party: Claudia Walther, University of Leipzig, Department of Cardiology
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: Leipzig aortic valve study
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2010-01-14 (Estimated); Status verified 2006-09

CONDITIONS: Aortic Valve Stenosis
Keywords: aortic valve stenosis; statin therapy
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — Fluvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

INTERVENTIONS:
Drug: fluvastatin — 40mg fluvastatin daily

SUMMARY:
There is evidence that the degenerative changes leading to aortic stenosis are caused by a chronic inflammatory process. Furthermore the development of aortic stenosis is partially dependent on typical cardiovascular risk factors. An inflammatory process as well as those risk factors are amenable for medical therapy. As such the use of statins (HMG CoA reductase inhibitors) would be an appealing concept to reduce both those risks for development of aortic stenosis. Aim of this study is to evaluate the usefulness of statin therapy on the progression of aortic stenosis.

DETAILED DESCRIPTION:
This study will be a prospective, double-blind, placebo-controlled, two-armed clinical trial trial to test the influence of statin therapy on the progression of calcified aortic stenosis in patients with asymptomatic mild to moderate aortic stenosis. After completion of all baseline investigations patients will be randomly assigned to the verum group (fluvastatin group) or to the control group (placebo group). Patients in the verum group will receive fluvastatin in a starting dose of 40 mg per day. The dose should be increased up to 80 mg per day. The treatment should be continued until the study end (24 months). Follow up investigations will be performed after 6, 12, and 18 months. After 24 months the final investigations will be performed.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 21 years
2. Mild to moderate aortic stenosis
3. No symptoms caused by aortic stenosis
4. Written informed consent to participate in the study
5. Aortic valve leaflet thickening with reduced systolic opening
6. Reduced aortic valve area > 0,8 cm2 and < 1,5 cm2
7. Maximum aortic jet velocity at rest > 2,5 m/s

Exclusion Criteria:

1. Symptoms caused by aortic stenosis
2. Aortic valve area < 0,7 cm2
3. Severe aortic regurgitation
4. Reduced left ventricular ejection fraction (< 50%)
5. Any valve disease with indication for surgery
6. Coronary artery disease
7. Therapy refractory arterial hypertension
8. Comorbid noncardiac diseases or other reasons which make a regular follow-up impossible
9. Other indication for treatment with statins
10. Women of childbearing potential not using the contraception method(s) specified in this study (specify), as well as women who are breastfeeding
11. Known sensitivity to study drug(s) or class of study drug(s)
12. Patients with severe medical condition(s) that in the view of the investigator prohibits participation in the study (specify as required)
13. Use of any other investigational agent in the last 30 days

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2003-01; Primary Completion 2009-09 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Progression of calcified aortic stenosis measured by: | 24 months
Transthoracic echocardiography (P max/ mean; V max; AVA) | 24 months
Catheterization (peak to peak gradient, LV-function, compliance) | 24 months

SECONDARY OUTCOMES:
Number of cardiovascular events | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Schuler, Professor, Principal Investigator
Locations (1):
- University of Leipzig - Heart Center, Leipzig, Saxony, Germany